CLINICAL TRIAL: NCT05927896
Title: Reliability and Validity of the Turkish Version of the 6-item Carpal Tunnel Syndrome Symptoms Scale
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Sezin Solum, MD; Physical Medicine & Rehabilitation Specialist Physician, Bursa City Hospital
Other Study IDs: 9999999991
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome; Symptoms and Signs
Keywords: carpal tunnel syndrome; Boston Carpal Tunnel Questionnaire; validity; Turkish adaptation; reliability; 6-item Carpal Tunnel Syndrome Symptoms Scale
MeSH Terms: conditions — Carpal Tunnel Syndrome; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 6-item Carpal Tunnel Syndrome Symptoms Scale — 6-item Carpal Tunnel Syndrome Symptoms Scale is a self-reported 6 item questionnaire.

SUMMARY:
Carpal tunnel syndrome (CTS) is a common condition that affects the median nerve that usually cause numbness, tingling, pain, and weakness in the hand and fingers. While definitive diagnosis is made with nerve conduction studies, the patient's history and physical examination findings lead the clinician to the diagnosis of CTS. Using factor analysis and item response theory methodology, Atroshi et al. developed a short 6-item version of the symptom severity scale to ease respondent burden while maintaining the psychometric properties of the Boston Carpal Tunnel Questionnaire. It has been demonstrated that the 6-item CTS Symptom Scale has good reliability, validity and responsiveness.

The aim of this study was to evaluate the reliability and construct validity of the Turkish version of the 6-item CTS symptoms scale for CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common condition that affects the median nerve that usually cause numbness, tingling, pain, and weakness in the hand and fingers. While definitive diagnosis is made with nerve conduction studies, the patient's history and physical examination findings lead the clinician to the diagnosis of CTS. The use of patient-completed disease-specific scales is increasing in clinical research and patient follow-up. Various scales have been developed to question symptoms related to hand problems. The Boston Carpal Tunnel Questionnaire and the 6-item CTS Symptom Scale are the scales that have been shown to be used to assess symptom severity and for diagnostic screening. Using factor analysis and item response theory methodology, Atroshi et al. developed a short 6-item version of the symptom severity scale to ease respondent burden while maintaining the psychometric properties of the Boston Carpal Tunnel Questionnaire . It has been demonstrated that the 6-item CTS Symptom Scale has good reliability, validity and responsiveness.

The aim of this study was to evaluate the reliability and construct validity of the Turkish version of the 6-item CTS symptoms scale for CTS.

ELIGIBILITY:
Inclusion Criteria:

* presence of numbness or tingling in at least two radial side fingers,
* a positive Phalen's test result,
* symptoms lasting more than three months
* consistent nerve conduction study with CTS.

Exclusion Criteria:

* those with no electrophysiological evidence of CTS,
* diabetes or other metabolic diseases,
* any other inflammatory diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 Carpal Tunnel Syndrome patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
6-item CTS Symptom Scale (CTS-6) | baseline
  The CTS-6 is a scale designed to measure the severity of CTS symptoms. It consists of six items, five of which are similar to those on the symptom severity subscale of the Boston CTS Scale, while the sixth item is a combination of two items from the same subscale.
Boston Carpal Tunnel Questionnaire (BCTQ) | baseline
  The BCTQ consists of two subscales, the Symptom Severity Scale and the Functional Status Scale. The Functional Status Scale contains eight items assessing activities such as "writing, buttoning clothes, holding a book while reading, grasping a telephone handle, opening a jar, doing housework, carrying grocery bags, bathing and dressing" whereas the 11-item Symptom Severity Scale assesses pain, paresthesia, numbness, weakness, nocturnal symptoms and grip difficulty.
The Michigan Hand Outcomes Questionnaire (MHQ) | baseline
  MHQ is a standardized instrument designed to quantify outcomes in patients with a range of hand conditions. The MHQ consists of 6 subscales: hand function, activities of daily living, pain, satisfaction, aesthetics and work performance. A cumulative score is calculated to provide an indication of overall function.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Salbaş, MD, Study Director — Balikesir University
Locations (1):
- Bursa Kestel State Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sevy JO, Sina RE, Varacallo MA. Carpal Tunnel Syndrome. 2023 Oct 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448179/ PMID 28846321
- [Background] Hoang-Kim A, Pegreffi F, Moroni A, Ladd A. Measuring wrist and hand function: common scales and checklists. Injury. 2011 Mar;42(3):253-8. doi: 10.1016/j.injury.2010.11.050. Epub 2010 Dec 15. PMID 21159335
- [Background] Chung KC, Pillsbury MS, Walters MR, Hayward RA. Reliability and validity testing of the Michigan Hand Outcomes Questionnaire. J Hand Surg Am. 1998 Jul;23(4):575-87. doi: 10.1016/S0363-5023(98)80042-7. PMID 9708370
- [Background] Schulze DG, Nilsen KB, Killingmo RM, Zwart JA, Grotle M. Clinical Utility of the 6-Item CTS, Boston-CTS, and Hand-Diagram for Carpal Tunnel Syndrome. Front Neurol. 2021 Jul 27;12:683807. doi: 10.3389/fneur.2021.683807. eCollection 2021. PMID 34385969
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Atroshi I, Lyren PE, Ornstein E, Gummesson C. The six-item CTS symptoms scale and palmar pain scale in carpal tunnel syndrome. J Hand Surg Am. 2011 May;36(5):788-94. doi: 10.1016/j.jhsa.2011.02.021. PMID 21527135
- [Background] Atroshi I, Lyren PE, Gummesson C. The 6-item CTS symptoms scale: a brief outcomes measure for carpal tunnel syndrome. Qual Life Res. 2009 Apr;18(3):347-58. doi: 10.1007/s11136-009-9449-3. Epub 2009 Feb 20. PMID 19229657
- [Background] Mollestam K, Rosales RS, Lyren PE, Atroshi I. Measuring symptoms severity in carpal tunnel syndrome: score agreement and responsiveness of the Atroshi-Lyren 6-item symptoms scale and the Boston symptom severity scale. Qual Life Res. 2022 May;31(5):1553-1560. doi: 10.1007/s11136-021-03039-1. Epub 2021 Nov 20. PMID 34800220
- [Background] Lyren PE, Atroshi I. Using item response theory improved responsiveness of patient-reported outcomes measures in carpal tunnel syndrome. J Clin Epidemiol. 2012 Mar;65(3):325-34. doi: 10.1016/j.jclinepi.2011.08.009. Epub 2011 Dec 15. PMID 22172153
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835